CLINICAL TRIAL: NCT02031965
Title: A Phase I Study of Intratumoral/Peritumoral Herpes Simplex Virus-1 Mutant HSV1716 in Patients With Refractory or Recurrent High Grade Gliomas (HGG)
Brief Title: Oncolytic HSV-1716 in Treating Younger Patients With Refractory or Recurrent High Grade Glioma That Can Be Removed By Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBTC-037; NCI-2013-00526 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-037 (Other: Pediatric Brain Tumor Consortium); PBTC-037 (Other: CTEP); U01CA081457 (NIH)
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Recurrent Childhood Anaplastic Astrocytoma; Recurrent Childhood Anaplastic Oligoastrocytoma; Recurrent Childhood Anaplastic Oligodendroglioma; Recurrent Childhood Giant Cell Glioblastoma; Recurrent Childhood Glioblastoma; Recurrent Childhood Gliomatosis Cerebri; Recurrent Childhood Gliosarcoma
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Neoplasms, Neuroepithelial | interventions — Dexamethasone; Calcium Dobesilate

ARMS (1):
- Treatment (oncolytic HSV-1716) (Experimental): Patients receive oncolytic HSV-1716 IT and peritumorally after undergoing surgical tumor resection. Patients also receive dexamethasone IV prior to and 6 and 12 hours after surgery.
  Interventions: Biological: oncolytic HSV-1716; Drug: dexamethasone; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: oncolytic HSV-1716 — Given IT
  Other Names: herpes simplex virus 1716
Drug: dexamethasone — Given IV
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Procedure: therapeutic conventional surgery — Undergo surgical resection
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and the safety of injecting HSV1716 (a new experimental therapy) into or near the tumor resection cavity. The injection will be done at the time of surgery. HSV1716 is a virus that has a gene which has been changed or removed (mutated) in such a way that lets the virus multiply in dividing cells of the tumor and kills the tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether intratumoral/peritumoral injection of HSV1716 (oncolytic HSV-1716) is safe in children with recurrent high-grade gliomas amenable to resection.

II. To estimate the maximum tolerated dose (MTD) or a recommended Phase II dose of intratumoral/peritumoral injection of HSV1716.

III. To describe any dose-limiting toxicities (DLT) of intratumoral/peritumoral injection of HSV1716 at the doses given to children with high-grade gliomas.

IV. To evaluate changes in tumor enhancement, quantitative magnetic resonance (MR) measures of tumor perfusion (relative cerebral blood volume [rCBV], transfer coefficient [k^trans], fractional blood-plasma volume [Vp] and extravascular extracellular space per unit volume tissue [Ve] values and apparent diffusion coefficient [ADC]) in response to HSV1716 injection.

SECONDARY OBJECTIVES:

I. To measure antiviral immune response in patients with refractory high-grade gliomas injected with HSV1716.

II. To measure the systemic viremia and viral shedding following intratumoral/peritumoral administration of HSV1716.

III. To preliminarily describe the antitumor activity of HSV1716 injection within the confines of a Phase I study.

IV. To evaluate anti-tumor immune cellular and humoral immune responses. V. To evaluate changes in fluorodeoxyglucose (FDG)- positron emission tomography (PET) uptake in response to HSV1716 injection.

VI. To evaluate changes in tumor choline values using magnetic resonance (MR) spectroscopy in response to HSV1716 injection and further delineate from progressive disease versus pseudo-progression post therapy.

OUTLINE: This is a dose-escalation study.

Patients receive oncolytic HSV-1716 intratumorally (IT) and peritumorally after undergoing surgical tumor resection. Patients also receive dexamethasone intravenously (IV) prior to and 6 and 12 hours after surgery.

After completion of study treatment, patients are followed up every 2 months for 1 year, every 6 months for 4 years, and then annually for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Imaging evaluations necessary to establish eligibility for study entry must be done within three (3) weeks prior to registration; all other evaluations necessary to establish eligibility for study entry must be done within two (2) weeks prior to registration; in the event that the patient's condition deteriorates (performance score < 60) within 48 hours prior to the injection the patient is no longer eligible to receive HSV1716 injection
* Patients must have a histologically-confirmed primary diagnosis of high-grade glioma (HGG) (such as glioblastoma multiforme, gliosarcoma, anaplastic oligodendroglioma, anaplastic ganglioglioma, high grade astrocytoma, not otherwise specified [NOS]) that is recurrent or refractory to conventional therapy; patients with metastatic disease are not eligible
* Patients must be those for whom surgical resection is clinically indicated; the intent of surgical resection may include debulking or attempt to resect as much of the tumor as safely feasible; if a gross total or near total resection is not feasible, HSV1716 injection into the wall of the resection cavity, encompassing residual tumor, is permissible

  * Patients must be amenable to receiving 1 dose of HSV1716 intra-operatively with planned HSV1716 injection sites >= 1 cm from the ventricular system AND meet at least one of the criteria below based upon pre-surgical magnetic resonance imaging (MRI):

    * Tumor is >= 1 cm from the ventricular system
    * Patients whose tumors that are =< 1 cm from the ventricular system are eligible if there is sufficient space within the tumor cavity and/or residual tumor to perform the HSV 1716 injections that are >= 1 cm from the ventricular system
  * An intraoperative MRI upon resection will confirm the distance of the planned injection sites from the ventricular system prior to the HSV1716 injection; intra-operatively, the neurosurgeon may decide to not inject the HSV1716 or may revise the sites of HSV1716 injection if injection cannot be guaranteed >= 1 cm from the ventricular system; patient will removed from the study if there are not sufficient areas in the tumor cavity to guarantee injection of HSV1716 >= 1 cm from the ventricular system
* Patients must have received prior therapy other than surgery and must have fully recovered from the acute treatment related toxicities of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study
* Patients must have received their last dose of known myelosuppressive anticancer chemotherapy at least three (3) weeks prior to study registration treatment or at least six (6) weeks if nitrosourea
* Investigational/Biologic agent:

  * Biologic or investigational agent (anti-neoplastic): Patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the investigational or biologic agent >= 7 days prior to study registration

    * For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur
  * Monoclonal antibody treatment: At least three half-lives must have elapsed prior to registration; Note: A list of the half-lives of commonly used monoclonal antibodies is available on the Pediatric Brain Tumor Consortium (PBTC) webpage under Generic Forms and Templates
* Patients must have had their last fraction of:

  * Craniospinal irradiation (> 24 Gray [Gy]) or total body irradiation > 3 months prior to registration
  * Focal irradiation to symptomatic metastatic sites > 4 weeks prior to registration
  * Local palliative external beam radiation therapy (XRT) (small port) >= 4 weeks
  * If prior total-body irradiation (TBI), craniospinal XRT or if >= 50% radiation of pelvis >= 6 months must have elapsed
  * If other substantial bone marrow (BM) radiation >= 6 weeks must have elapsed
* Patient must be:

  * >= 6 months since allogeneic bone marrow transplant prior to registration
  * Stem cell transplant or rescue without TBI: No evidence of active graft vs. host disease and >= 3 months must have elapsed since transplant
* Karnofsky performance scale (KPS for > 16 years of age) or Lansky performance score (LPS for =< 16 years of age) assessed within two weeks of registration must be >= 60
* Hemoglobin: >= 10 g/dl
* Absolute neutrophil count: >= 1000/mm^3
* Platelets: >= 100,000/mm^3 (transfusion independent defined as not receiving platelet transfusions within 7 days prior to registration)
* Total bilirubin: < 1.5 x upper limit of institutional normal for age
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]): =< 2.5 × institutional upper limit of normal
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age and gender as follows:

  * Age 10 to < 13 years: maximum serum creatinine (mg/dL): 1.2 for males and 1.2 for females
  * Age 13 to < 16 years: maximum serum creatinine (mg/dL): 1.5 for males and 1.4 for females
  * Age >= 16 years: maximum serum creatinine (mg/dL): 1.7 for males and 1.4 for females
* Albumin >= 2.5 g/dL
* Partial thromboplastin time (PTT) < 1.2 X institutional upper limits of normal
* Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to registration; this is to be documented at baseline
* Patients with central nervous system (CNS) tumors who are receiving dexamethasone must have been on a stable or decreasing dose of dexamethasone for the 7 days prior to enrollment
* Growth factors that support platelet or white cell number or function must not have been administered within the past 7 days; growth factors include: GCSF (filgrastim), PEG-GCSF (Neulasta), GM-CSF (sargramostim) and erythropoietin
* Documented evidence of negative tests for the presence of hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV)1/2 antibodies within the three months preceding study entry; subjects who do not have such evidence must undergo appropriate testing prior to virus administration; HIV-positive patients on combination antiretroviral therapy are ineligible
* Female patients of childbearing potential must have a negative serum or urine pregnancy test at the time of enrollment
* Ability to understand and the willingness to sign a written informed consent document according to institutional guidelines

Exclusion Criteria:

* Patients with metastatic disease i.e. leptomeninges, multi-focal lesions in the CNS
* Patients whose tumor lies within 1 cm of the ventricular system
* Patients who are receiving any other investigational agents
* Patients who are currently receiving other anti-cancer agents are excluded from this trial
* Patients with history of prior HSV encephalitis or encephalitis due to other etiologies
* There is no available information regarding human fetal or teratogenic toxicities
* Pregnant women are excluded to avoid the risk of systemic intrauterine/neonatal HSV infection
* Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method from the time of study entry to a period of no less than four months post the HSV1716 injection
* Women who participate in this study must agree not to breastfeed from study entry to a period of no less than four months post the HSV1716 injection
* Subjects whose primary physicians determine that anti-HSV antiviral therapy (such as acyclovir, ganciclovir, foscarnet, etc.) cannot be safely discontinued from 2 days prior to the injection to 28 days following the injection are excluded from this study
* Patients on systemic anticoagulants are excluded from this study
* Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that would compromise the patient's ability to tolerate protocol therapy or would likely interfere with the study procedures or results

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2013-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
MTD of oncolytic HSV-1716, defined as the highest dose level at which 0 out of 3 or at most one out of 6 patients have been treated experiencing a dose limiting toxicity and the next higher dose level has been determined to be too toxic | 56 days
  Graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0.

SECONDARY OUTCOMES:
Antiviral immune responses | Up to 15 years
  Summarized and reported descriptively.
Systemic viremia and viral shedding | Up to 15 years
  Summarized and reported descriptively.
Progression free survival | From the date of initial protocol treatment to the earliest date of disease progression, second malignancy or death for patients who fail; and to the date of last contact for patients who remain at risk for failure, assessed up to 15 years
Overall survival | From the date of initial protocol treatment to the date of death for patients who fail; and to the date of last contact for patients who remain at risk for failure, assessed up to 15 years
Changes in MR parameters (including diffusion and perfusion studies) (optional) | Baseline up to 2 months post-injection
  Summary statistics and graphs used to describe changes in these quantitative imaging parameters.
Changes in MRS and PET parameters (including diffusion and perfusion studies) (optional) | Baseline up to 2 months post-injection
  Summary statistics and graphs used to describe changes in these quantitative imaging parameters.
Anti-tumor cellular responses | Up to week 16
Humoral immune responses | Up to week 16

CONTACTS AND LOCATIONS:
Overall Officials: Mariko DeWire, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States